CLINICAL TRIAL: NCT07241039
Title: A Phase 1 First-in-Human, Open-Label Study Evaluating the Safety, Pharmacokinetics, and Efficacy of ABBV-711 as a Monotherapy or in Combination With Budigalimab (ABBV-181) in Adult Subjects With Advanced Squamous Tumors
Brief Title: A Study to Assess the Adverse Events, Change in Disease Activity, and How Oral ABBV-711 Tablets Move Through the Body as a Monotherapy and in Combination With Intravenously Infused Budigalimab (ABBV-181), in Adults With Advanced Squamous Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M25-632; 2025-521607-48-00 (Other: EU CT)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Advanced Squamous Tumors
Keywords: Advanced Squamous Tumors; ABBV-711; ABBV-181; Budigalimab; Head and Neck Squamous Cell Carcinoma; Squamous Non-Small Cell Lung Cancer; sqNSCLC; HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — budigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part 1: ABBV-711 Monotherapy Dose Escalation (Experimental): Participants will receive ABBV-711 in escalating doses alone, as part of the 5 year study duration.
  Interventions: Drug: ABBV-711
- Part 2a: ABBV-711 Monotherapy Dose Expansion (Experimental): Participants will receive ABBV-711 dose A alone, as part of the 5 year study duration.
  Interventions: Drug: ABBV-711
- Part 2b: ABBV-711 Monotherapy Dose Expansion (Experimental): Participants will receive ABBV-711 dose B alone, as part of the 5 year study duration.
  Interventions: Drug: ABBV-711
- Part 3: ABBV-711 + BudigalimabDose Escalation (Experimental): Participants will receive ABBV-711 in escalating doses in combination with budigalimab, as part of the 5 year study duration.
  Interventions: Drug: ABBV-711; Drug: Budigalimab
- Part 4a: ABBV-711 Budigalimab Dose Expansion (Experimental): Participants will receive ABBV-711 dose A in combination with budigalimab, as part of the 5 year study duration.
  Interventions: Drug: ABBV-711; Drug: Budigalimab
- Part 4b: ABBV-711 Budigalimab Dose Expansion (Experimental): Participants will receive ABBV-711 dose B in combination with budigalimab, as part of the 5 year study duration.
  Interventions: Drug: ABBV-711; Drug: Budigalimab

INTERVENTIONS:
Drug: ABBV-711 — Oral Tablet
Drug: Budigalimab — Intravenous Infusion
  Arms: Part 3: ABBV-711 + BudigalimabDose Escalation; Part 4a: ABBV-711 Budigalimab Dose Expansion; Part 4b: ABBV-711 Budigalimab Dose Expansion

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. The purpose of this study is to assess safety, tolerability, pharmacokinetics and preliminary efficacy of ABBV-711 as a monotherapy and in combination with budigalimab (ABBV-181) in adults with advanced squamous tumors.

ABBV-711 is an investigational drug being developed for the treatment of solid tumors. There are multiple treatment arms in this study. Participants will either receive ABBV-711 as a single agent or in combination with budigalimab (another investigational drug) at different doses. Approximately 220 adult participants will be enrolled in the study across 40 sites worldwide.

In part 1, oral ABBV-711 tablets will be given in escalating doses alone to participants with squamous (sq) tumors. In part 2 oral ABBV-711 tablets will be given at a selected dose from part 1 to participants with squamous non-small cell lung cancer (sqNSCLC), or head and neck squamous cell carcinoma (HNSCC). In part 3, oral ABBV-711 tablets will be given in escalating doses in combination with intravenously (IV) infused budigalimab to participants with sq tumors. In part 4 oral ABBV-711 tablets will be given at a selected dose from part 3 in combination with IV infused budigalimab to participants with sqNSCLC, or HNSCC. The estimated duration of the study is up to approximately 5 years.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent questionnaire, medical assessments, blood tests, and scans.

ELIGIBILITY:
Inclusion Criteria:

* Must have progressed on or after standard of care therapy and have no curative therapy available (participants who have refused, are considered ineligible for or are intolerant to standard of care therapy are eligible).
* Received programmed cell death protein 1 (PD-1)/programmed cell death ligand 1 (PD-L1) targeted agents are eligible.
* Confirmation of available archival tumor tissue (formalin-fixed paraffin-embedded [FFPE] block or freshly cut slides) or provision of fresh tissue biopsy is required for enrollment in this study for gene expression assessment. If archival tissue requirements cannot be met then the AbbVie therapeutic area Medical Director or designee should be contacted to determine subject eligibility.
* For head and neck squamous cell carcinoma (HNSCC) participants enrolled in backfill (Part 1 and 3), subjects must provide consent to paired biopsies which are pretreatment and on treatment fresh tumor biopsies from the same tumor lesion, unless deemed not feasible by the investigator where upon consultation with the Sponsor is required. Paired biopsies are encouraged (when safe and feasible) but not required for subjects with squamous non-small cell lung cancer (sqNSCLC) enrolled in the backfill (Part 1 and 3).
* Evaluable and measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.

Exclusion Criteria:

* Active autoimmune diseases besides vitiligo, type 1 diabetes, hypothyroidism, hypopituitarism and psoriasis (not requiring systemic treatment); history of primary immunodeficiency, bone marrow transplantation, or solid organ transplantation. Active inflammatory bowel disease unfit for trial in the opinion of the investigator, including subjects requiring systemic therapy with biologics or immunosuppressive therapy within the past 2 years.
* Treatment with any of the following:

  * Anti-cancer therapy including chemotherapy, radiation therapy, immunotherapy, biologic, or any investigational therapy within 28 days or 5 half-lives of the drug (whichever is shorter) prior to the first dose of ABBV-711. Palliative radiation therapy for bone, skin or symptomatic metastases with 10 fractions or less is not subject to a washout period.
  * Radiation therapy for central nervous system metastases within 14 days prior to first dose.
* Subject has systemically used known moderate/strong inhibitors of cytochrome P450 3A (CYP)3A enzyme isoform subfamily within 14 days or 5 half-lives of the drug (whichever is shorter) prior to the first dose of study treatment.
* Has systemically used known moderate/strong inducers of CYP3A within 14 days prior to the first dose of study treatment.
* Requires treatment with known moderate or strong inhibitors or inducers of CYP3A from the first dose of study treatment and for the duration of the study.
* Administration or consumption of any of the following within 3 days prior to first dose of study treatment and while on study treatment: grapefruit or grapefruit products, Seville oranges (including marmaladecontaining Seville oranges), and star fruit.
* Current or prior use of immunosuppressive medication within 14 days prior to the first dose of the study treatment. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids or local steroid injections (e.g., intra-articular injection);
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication);
  * Systemic corticosteroids at doses not to exceed 10 mg/day of prednisone or equivalent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE)s | Up to Approximately 5 Years
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Best overall Response (BOR) | Up to Approximately 5 Years
  BOR is defined as partial response (PR) or better per investigator review according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Duration of BOR Response | Up to Approximately 5 Years
  Duration of response for participants with confirmed PR or better.
Clinical Benefit Rate (CBR) | Up to Approximately 5 Years
  CBR is defined as the percentage of participants with BOR of stable disease (SD) or BOR of PR or better per investigator review according to RECIST version 1.1 criteria.
Progression-free survival (PFS) | Up to Approximately 5 Years
  PFS is defined as time from first ABBV-711 to a documented disease progression according to RECIST version 1.1, as determined by the investigator, or death due to any cause, whichever occurs earlier.
Duration of response (DOR) | Up to Approximately 5 Years
  DOR is defined for participants achieving a confirmed PR or better as the time from the initial response of PR (or better) per investigator review according to RECIST 1.1 or other criteria to disease progression or death of any cause, whichever occurs earlier.
Overall survival (OS) | Up to Approximately 5 Years
  OS is defined as time from first ABBV-711 to death due to any cause.
Area Under the Concentration-Time Curve (AUC) of ABBV-711 | Up to Approximately 5 Years
  Area under the concentration-time curve of ABBV-711.
Maximum Observed Concentration (Cmax) of ABBV-711 | Up to Approximately 5 Years
  Maximum observed concentration of ABBV-711.
Time to Cmax (Tmax) of ABBV-711 | Up to Approximately 5 Years
  Time to Cmax of ABBV-711.
Half-Life (t1/2) of ABBV-711 | Up to Approximately 5 Years
  Half-life of ABBV-711.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (7):
- United States (3):
  - START Midwest /ID# 272505, Grand Rapids, Michigan
  - Carolina BioOncology Institute /ID# 272380, Huntersville, North Carolina
  - Next Oncology - Irving /ID# 276659, Irving, Texas
- Israel (3):
  - The Chaim Sheba Medical Center /ID# 276798, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus /ID# 276799, Haifa
  - Hadassah Medical Center-Hebrew University /ID# 276800, Jerusalem
- Kansai Medical University Hospital /ID# 276586, Hirakata-shi, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-632